CLINICAL TRIAL: NCT02152436
Title: Simulation-based Curriculum to Enhance Culture of Safety in Operating Rooms
Acronym: PROPECS
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-32
Record Dates: First submitted 2014-03-20; First posted 2014-06-02 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before simulation-based curriculum: 125 surgical interventions will be observed and outcomes will be measured before simulation-based curriculum
- After simulation-based curriculum: 125 surgical interventions will be observed and outcomes will be measured after simulation-based curriculum
  Interventions: Other: Simulation - based curriculum

INTERVENTIONS:
Other: Simulation - based curriculum — Operating room medical and non-medical members will be asked to carry out a simulation session preceded by an educational maze with videos. Outcomes will be compared and correlated after and before this curriculum
  Groups: After simulation-based curriculum

SUMMARY:
Communication in the operating room (OR) is a key factor to prevent deleterious events for the patient. French national health authority made the implementation of safety checklist mandatory in operating rooms. The goal of this checklist is to improve teamwork and share key elements for better patient outcomes. Observational studies in the OR showed low compliance to this checklist, either on the way it is used or on the information implemented.

The primary objective of this project is to assess the efficacy of a simulation-based curriculum involving OR medical and non-medical personnel in order to improve communication in the OR.

DETAILED DESCRIPTION:
Operating theater is a complex system where efficient communication is critical to patient safety. Patient safety check-list are used worldwide as a way to improve communication and teamwork in the operating room in order to decrease perioperative morbidity and mortality. Previous studies have shown that communication failure in the OR may be associated with adverse events. The improvement of safety culture (including communication and team work) may be obtained by simulation based training.

The primary objective of this before-after study is to assess the efficacy of a simulation-based curriculum involving OR medical and non medical personnel in order to improve communication in the OR.

In brief, in a first period, an audit to assess communication efficacy and teamwork will be realized during 125 surgical procedures. Communication failures and consequences will be recorded using a standardized form filled by trained personnel. In a second phase, all the OR personnel (surgeon, anesthesiologist, nurses) will be invited to participate to a special training on communication and teamwork. This curriculum will include formal presentations and also simulation-based training. Scenarios are built to improve the ability to communicate in specific situations (fire in the OR, haemorrhage, wrong side, anaphylaxis).

In a third phase, an audit on communication and teamwork, similar to the first phase will be realized. The primary endpoint is the frequency of surgical interventions having at least one communication failure with a consequence. The investigators expect a significant decrease in the rate of communication failures between phase 1 and 3. A fourth phase will consist in a last audit two years after phase 1 to evaluate long-term effect of this curriculum.

ELIGIBILITY:
Inclusion Criteria:

* All surgical interventions occuring in Grenoble University Hospital, North site, between November and January

Exclusion Criteria:

* Interventions supposed to last more than 4 hours
* Interventions in situations of vital emergencies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgical interventions in Grenoble University Hospital
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Frequency of surgical interventions having at least on communication failure with a consequence | After 3 months of audit

SECONDARY OUTCOMES:
Compliance to the safety checklist in the operating room | measured during each surgical intervention, before anesthesia, before incision and at the end of surgery
6 items survey estimating teamwork quality | measured at the end of each surgical intervention, an average of 2.5 hours
Number of adverse events occuring in the OR declared to the institution | After 3 months of audit
Surgical Apgar score | measured at the end of each surgical intervention, an average of 2.5 hours
Nature of communication failure and consequences | measured during each surgical procedure, for an average of 2.5 hours
rate of communication failures | measured during each surgical procedure, for an average of 2.5 hours
Survey on safety culture for employees working in the OR | After 3 months of audit
Count of team members and number of passage in the OR | measured during each surgical procedure, for an average of 2.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Albaladejo, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Operating rooms of Grenoble University Hospital, Grenoble, France